CLINICAL TRIAL: NCT03464474
Title: Evaluation of Digital Holographic Microscopy for Quantification and Characterization of the Histological Disease Activity in Patients With Ulcerative Colitis
Brief Title: Digital Holographic Microscopy: Evaluation of Histological Disease Activity in Patients With Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-476-f-S
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Quantitative Phase Imaging

STUDY DESIGN:
Intervention Model Description: Colonic biopsies from 28 patients with ulcerative colitis will be endoscopically acquired. These biopsies will be examined by digital holographic microscopic and by analysis due to an experienced histopathologists using an established scoring system (Goldstandard).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of inflammation grade (Experimental): Colonic biopsies will be acquired. Biopsies from all patients will be examined using digital holographic microscopy as well as performing a histopathological analysis using the Nancy-score (Goldstandard).
  Interventions: Device: digital holographic microscopy

INTERVENTIONS:
Device: digital holographic microscopy — Colonic biopsies from all patients will be assessed using digital holographic microscopy in comparison to the existing Goldstandard (histopathological analysis).

SUMMARY:
Ulcerative colitis (UC) belongs to the group of inflammatory bowel disease (IBD) and is characterized by a chronic relapsing disease course. As uncontrolled intestinal inflammation can lead to severe disease complications, treatment of UC has evolved from sole treatment of symptoms up to histological remission which is marked by the absence of histological inflammation. To correctly assess and quantify the degree of histological inflammation in IBD patients remains difficult.

Digital holographic microscopy (DHM) is a new imaging technique belonging to quantitative phase contrast imaging. It is based on the detection of optical path-length delays in a stain-free manner, thereby providing a refractive index which directly correlates to tissue density.

This study aims to evaluate the role of DHM for quantifying the degree of histological inflammation in endoscopically acquired biopsies of UC patients in a prospective clinical trial. From 28 UC patients, the investigators will obtain endoscopically acquired colonic biopsies. The investigators will assess the degree of inflammation in these biopsies using DHM and in addition to this an experienced histopathologist will determine the degree of inflammation in these biopsies using a histological scoring system (Nancy-Score = goldstandard). Finally, the investigators will directly correlate the results from DHM analysis to the histological analysis using the Nancy-Score.

ELIGIBILITY:
Inclusion Criteria:

- Patients with an indication for a colonoscopy

Exclusion Criteria:

* Patients under 18 years, pregnancy
* Inability to have a patient education
* Bad conditions or other reasons prohibiting a colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of the inflammation grade of mucosal biopsies of ulcerative colitis patients | Endoscopically acquired biopsies will immediately be transported to the laboratory. After processing, biopsies can be used for histological assessment and for digital holographic microscopy; biopsies will be assessed within a time period up to 56 weeks.
  From patients with ulcerative colitis, the investigators will collect endoscopically acquired colonic biopsies. For the primary outcome, the investigators will correlate the conventional histological analysis using an established histological scoring system (Nancy-Score) in comparison to the experimental procedure using digital holographic microscopy thereby determining a refractive index which directly correlates to tissue density.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Bettenworth, Professor, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Unversity Clinic Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided